CLINICAL TRIAL: NCT01878968
Title: Does Detailed Informed Consent for Cardiopulmonary Resuscitation and Mechanical Ventilation Impact Patients' Decisions and Outcomes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish Hospital, Cincinnati, Ohio (Other)
Responsible Party: Principal Investigator, Imran Naqvi, Chief Hospitalist, Associate Program Director Internal Medicine Residency, Jewish Hospital, Cincinnati, Ohio
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-06
Record Dates: First submitted 2013-05-07; First posted 2013-06-17 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Congestive Heart Failure; Infections; Sepsis; Acute Renal Failure; Stroke
MeSH Terms: conditions — Heart Failure; Infections; Sepsis; Acute Kidney Injury; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Script and Video (Experimental): Patients in the Script and CPR/Mechanical ventilation video arm will receive information on CPR and mechanical ventilation via a script and a video.
  Interventions: Other: Script and CPR/Mechanical ventilation video.
- Script only (Experimental): Patients in the Script only arm will receive information on CPR and mechanical ventilation via a script only.
  Interventions: Other: Script and CPR/Mechanical ventilation video.

INTERVENTIONS:
Other: Script and CPR/Mechanical ventilation video. — Patients will be randomized to receive the script (see addendum) plus video. Video was produced by and is the property of the study investigators.

SUMMARY:
There is evidence to suggest that patients make different end-of-life decisions if they understand the risks, benefits and alternatives of CPR and mechanical ventilation. This study will examine whether evidence-based informed consent impacts patients choices and healthcare outcomes compared to routine care.

ELIGIBILITY:
Inclusion Criteria:

* All patients
* ≥65 yrs
* Admitted to the hospitalist Medicine Service

Exclusion Criteria:

* Patients who have pre-existing, pan-institutional (e.g. to be applied at nursing homes and hospitals) orders of no CPR and/or no mechanical ventilation will be screened (demographic and outcomes data collected) but NOT randomized.
* Patients already receiving critical care on admission will also be excluded

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of patients opting out of routine care - no intubation | 48 hours
  Number of patients in each group who opt out of intubation 48 hours after admission.
Number of patients opting out of routine care - no CPR | 48 hours
  Number of patients in each group who opt out of CPR within 48 hours of admission.

SECONDARY OUTCOMES:
Hospital Mortality | Length of patient's hospital stay
  Number of deaths in each group in the hospital
30-day mortality | 30 days
  Number of deaths in each group after 30 days.
90 day mortality | 90 days
  Number of deaths in each group in 90 days.
Number of patients undergoing CPR | Length of patient's hospital stay
  Number of patients in each group who undergo CPR during their hospitalization.
Number of patients undergoing intubation | Length of patient's hospital stay
  Number of patients in each group who undergo intubation during their hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Naqvi, MD, Principal Investigator — Jewish Hospital of Cincinnati
Locations (1):
- The Jewish Hospital, Cincinnati, Ohio, United States